CLINICAL TRIAL: NCT06063330
Title: A Phase 1, Multicenter, Randomized, Double-blind, Placebo- Controlled, Parallel Group Study to Evaluate the Safety of RQ-01 in SARS-CoV-2 Positive Subjects
Brief Title: Clinical Trial to Evaluate the Safety of RQ-01 in SARS-CoV-2 Positive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Red Queen Therapeutics, Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RQ-01-001
Record Dates: First submitted 2023-09-17; First posted 2023-10-02 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: COVID-19; Infectious Disease; Symptomatic COVID-19 Infection Laboratory-Confirmed; SARS CoV 2 Infection
Keywords: First in Human; Phase 1; COVID; Telemedicine
MeSH Terms: conditions — COVID-19; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: There are 3 different treatment arms that subjects will be randomized in a 1:1:1 ratio. The arms will be evenly distributed with 22 subjects in each arm: 1) low dose of RQ-01; 2) high dose of RQ-01; 3) Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Low Dose of RQ-01 (Experimental): Subjects in this arm will receive 5 mg per day (for 3 days) of RQ-01
  Interventions: Combination Product: RQ-001
- High Dose of RQ-01 (Experimental): Subjects in this arm will receive 10 mg per day (for 3 days) of RQ-01
  Interventions: Combination Product: RQ-001
- Placebo (Placebo Comparator): Subjects in this arm will receive 0 mg per day (for 3 days) of RQ-01
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: RQ-001 — Drug product RQ-001 is the fully assembled device consisting of the vial containing RQ-01 and the actuator. Drug Product RQ-001 has been developed with an Aptar Bidose liquid nasal spray unit device (BDSI V3) capable of intranasally delivering a 200 uL total volume of drug product (specifically, 100 uL per nare, which delivers a 200 uL of total volume). The combination product comprises the drug constituent (RQ-01) and the assembly of commercially available, off-the-shelf device components.
  Study staff will be responsible for assembling the drug product RQ-001 and subjects will self-administer under the supervision of study staff in the clinic.
  Arms: High Dose of RQ-01; Low Dose of RQ-01
Other: Placebo — Matching placebo will be manufactured just as RQ-01 drug substance, with the active ingredient addition step omitted. Placebo will appear similar to RQ-01 drug substance as a clear to hazy, colorless to yellowish liquid. Matching placebo will be administered the same way as RQ-01
  Arms: Placebo

SUMMARY:
This is a first in human clinical study to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of RQ-01. Adult patients who have tested positive for SARS-CoV-2 virus, have mild symptom(s) of COVID-19 disease, and who are at low risk for developing moderate or severe COVID-19 disease are welcome to participate. The main questions this study aims to answer are:

1. What is the safety profile of RQ-01?
2. What is the reduction in SARS-CoV-2 ribonucleic acid (RNA) shedding after administration of RQ-01?
3. How effective is RQ-01 versus placebo in reducing COVID-19 symptoms?

After providing informed consent, subjects will be randomized to RQ-01 (high or low dose) or placebo and will be dosed for 3 consecutive days. Throughout the duration of the trial, subjects will participate in the following activities: perform rapid antigen and polymerase chain reaction (PCR) tests for COVID-19, answer questions about their medical history and medications, answer questions about their COVID-19 history and symptoms, conduct a physical exam, have their vitals measured, and have bloodwork done.

DETAILED DESCRIPTION:
This is a first in human study to evaluate the safety, PK, and PD of RQ-01 when administered to adult subjects who have tested positive for SARS-CoV-2 virus, have mild symptom(s) of COVID-19 disease, and who are at low risk for developing moderate or severe COVID-19 disease. Subjects will be exposed to RQ-01 after nasal administration with the Aptar Bidose nasal spray device (BDSI V3). The decrease in SARS-CoV-2 RNA shedding will be measured by reverse transcription-quantitative polymerase chain reaction (RT- qPCR) compared with placebo. There are currently no Food and Drug Administration (FDA) approved therapies for subjects with mild symptoms of COVID who are low risk for progression to moderate-severe disease. Safety of the subjects in this study is supported by the safety margin for local adverse events, lack of systemic exposure, and availability of antiviral therapies for COVID-19 should subjects' disease progress.

The study may be conducted using traditional outpatient clinic sites or a hybrid model, using clinic sites and/or virtual sites, with provisions made to conduct aspects of the study via telehealth and/or within subjects' homes. The hybrid model will provide the flexibility required to offer the trial in areas with increased incidence of COVID-19 disease, to maximize access to trial participation, and to increase diversity of trial subjects.

Potential study subjects will be identified for screening based on having at least one mild symptom consistent with COVID-19 disease. Potential study subjects may additionally present with a positive SARS-CoV-2 rapid antigen test (RAT), taken either at-home, or administered at a facility (e.g., urgent care testing site). As detailed within the inclusion criteria, different entry requirements apply depending on the source and timing of the positive rapid antigen test. For all subjects, the time from first positive SARS-CoV-2 rapid antigen test result to time of first dose must not exceed 3 days. Also, the first dose of study drug must be administered within 4 days of the estimated initial onset of symptoms of COVID-19 disease.

Subjects who provide written informed consent and meet all eligibility criteria will be randomized in a 1:1:1 manner to RQ-01 (high or low dose) or placebo. On the day of randomization, all subjects must have at least one mild symptom of COVID-19 disease and a positive SARS-CoV-2 RAT result. After the first six subjects are enrolled (2 in each group) and have completed all study procedures through Day 7 an early interim safety analysis will be performed by the Data Monitoring Committee. Enrollment of new subjects will continue only after review by the Data Monitoring Committee and the decision to proceed communicated to the investigators.

Prior to the first dose of study drug, all subjects must be trained by study staff on study drug self-administration with the Aptar Bidose nasal spray device, per the instructions provided within the Pharmacy Manual and/or subject-facing materials. Subjects will self-administer all doses of study drug while observed in-person by the Investigator or designee, who must be a trained healthcare professional. Subjects will then be followed for an additional 30 days for overall safety including COVID-19 disease symptoms.

If at any point during the study a subject meets the treatment discontinuation criteria outlined within the protocol, including a worsening of COVID-19 disease symptoms, the subject will be immediately discontinued from study drug and will continue in follow-up as described within the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64, inclusive, at the time of consent.
* Have mild COVID-19 disease symptom(s) at screening and at randomization, as defined in the protocol.
* Female subjects must have a negative urine pregnancy test at screening.
* Females of childbearing potential must agree to abstain from heterosexual intercourse or use highly effective contraception, as defined in the protocol.
* Male subjects must agree to abstain from heterosexual intercourse or use double barrier protection with condom and spermicide with any sexual partner who has the capacity for pregnancy and agree to not donate sperm.
* Understand the risks of the trial and consents to study conduct documented by signing of the study informed consent form.
* Willing and able to comply with this protocol and be available for the entire duration of the study.

Exclusion Criteria:

* Moderate or severe COVID-19 disease at the time of screening, including but not limited to displaying one or more of the following clinical symptoms outlined in the protocol
* Individuals who are eligible for FDA authorized or approved COVID-19 therapeutics (e.g., antivirals or monoclonal antibodies)
* Subjects at high-risk for COVID-19 disease severity progression at the time of screening, defined as subjects with known history or current diagnoses of any of the following conditions outlined in the protocol.
* Sinusitis ongoing for more than 4 weeks at the time of screening.
* Clinically significant epistaxis, as determined by the Investigator, within 3 months prior to screening.
* Nasal or sinus surgery within 12 weeks prior to screening, planned to occur during the study, or a history of any nasal or sinus surgery that in the opinion of the Investigator may influence COVID-19 disease symptoms or spray administration of the study drug.
* Nasal polyps or other non-infectious condition that could cause nasal obstruction, such as severe nasal septal deviation.
* Use of intranasal, inhaled, or oral corticosteroid medications of any kind within 14 days prior to the first dose of study drug, or planned use during the study that may affect the administration and/or absorption of study drug. Note: The use of oral antihistamines is permitted during the study.
* Use of antivirals or monoclonal antibodies for the management of COVID-19 disease or other viruses (e.g., influenza) within 60 days prior to the first dose of study drug.
* Received a vaccination for COVID-19 disease (original series or boosters) within 30 days prior to the first dose of study drug, and/or has plans to receive a COVID-19 vaccination (original series or boosters) during the trial through Day 33. Note: Other vaccinations are permitted during the trial through Day 33 and must be reported as a concomitant treatment.
* Have known systemic hypersensitivity to the RQ-01 drug substance, its inactive ingredients, or the ingredients of the matching placebo.
* For female subjects, are pregnant or breastfeeding, are < 1 month post-partum or are planning to become pregnant during the study.
* Have any condition that, in the opinion of the Investigator, would interfere with evaluation of the study drug or interpretation of the subject's safety or study results.
* Unwilling to abstain from participating in another interventional clinical study with an investigational compound or device, including SARS-CoV-2 therapeutics.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Incidence of TEAEs | Through 33 days
  The difference between treatment arms in the incidence of treatment-emergent adverse events (TEAEs) leading to withdrawal of study drug or study discontinuation through Day 33/End of Study.
Change in clinical laboratory results | Through 33 days
  The difference between treatment arms in the change from baseline in clinical laboratory results.
Change in physical examination results | Up to 33 days
  The difference between treatment arms in the change from baseline in physical examination results.
Change in vital signs | Up to 33 days
  The difference between treatment arms in the change from baseline in vital signs.

SECONDARY OUTCOMES:
Change in SARS-CoV-2 RNA shedding | Through 33 days
  The difference between treatment arms in the time-weighted average change in log10 SARS-CoV-2 SARS-CoV-2 RNA shedding from Baseline (Day 1) through Day 33 as measured by RT-qPCR.
Proportion of subjects with undetectable SARS-CoV-2 RNA shedding | Up to 33 days
  The difference between treatment arms in the proportion of subjects with undetectable SARS-CoV-2 RNA shedding as measured by RT-qPCR by visit.
Change in SARS-CoV-2 RNA shedding | Up to 5 days
  The difference in the change from baseline to Day 5 between treatment arms in the AUC SARS-CoV-2 RNA shedding as measured by RT-qPCR.
Proportion of subjects with negative RT-qPCR | Through 33 days
  The difference between treatment arms in the proportion of subjects with negative RT-qPCR through Day 33.
Time to negative RT-qPCR | Up to 33 days
  The difference between treatment arms in the time to negative RT-qPCR.
Proportion of rebounds | Through 33 days
  The difference between treatment arms in the proportion of rebounds (defined as: viral RNA ≥lower limit of quantitation (LLOQ) after Day 5 if <LLOQ at Day 5, or ≥1 log10 increase in viral RNA copy number (relative to Day 5) after Day 5 if ≥LLOQ at Day 5.
Proportion of subjects using additional therapeutic alternatives | Through 33 days
  The difference in proportion between treatment arms of subjects who used additional therapeutic alternatives for the management COVID-19 disease (as recommended by the National Institutes of Health [NIH]) for non-hospitalized COVID-19 subjects by treatment arms through Day 33.
Proportion of subjects with no symptoms | Through 33 days
  The difference in proportion between treatment arms of subjects with no symptoms through Day 33 as measured by the 15 items COVID-19 Symptoms Score.
Mean change in symptoms | Through 33 days
  The difference in the mean change from baseline through Day 33 as measured by the 15 items COVID-19 Symptoms Score.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Eisenberg, MD, MPH, Study Director — Red Queen Therapeutics
Locations (6):
- United States (6):
  - LA Universal Research Center, Inc., Los Angeles, California
  - Florida International Medical Research, Miami, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Zenos Clinical Research, Dallas, Texas
  - Vilo Research Group, L.L.C., Houston, Texas
  - Evergreen Hospital Medical Center, Kirkland, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — https://www.movecovidmedicineforward.com